CLINICAL TRIAL: NCT06445790
Title: Efficacy of Cognitive Behavior Therapy in the Treatment of Chronic Pelvic Pain in Women: A Randomized Controlled Trial
Brief Title: Efficacy of Cognitive Behavior Therapy in the Treatment of Chronic Pelvic Pain in Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Islamia University of Bahawalpur (Other)
Responsible Party: Principal Investigator, Bushra Akram, PhD Scholar, Islamia University of Bahawalpur
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUB
Record Dates: First submitted 2024-03-29; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pelvic Pain Syndrome
Keywords: Chronic Pelvic Pain, Pelvic Pain, Women
MeSH Terms: conditions — Pelvic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): It will receive 12 sessions of Cognitive Behavior Therapy for Chronic Pelvic Pain.
  Interventions: Behavioral: Cognitive Behavior Therapy for Chronic Pelvic Pain-CBT-cp
- Group B (No Intervention): Group B will be control group.

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy for Chronic Pelvic Pain-CBT-cp — CBT-cp will be administered weekly sessions for 12 weeks.
  Arms: Group A

SUMMARY:
This will be the pilot study trial. The target population will be 30 individuals with Chronic Pelvic Pain (CCP). There will be 02 groups, Experimental Group and Control Group. The primary outcome measure will be Impact of Female Chronic Pelvic Pain Questionnaire (IF-CPPQ). The experimental group will receive CBT spread over 12 sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Women of reproductive age.
2. Women with Chronic Pelvic Pain having no pathological or anatomical causes.
3. Women with Overactive Bladder Syndrome.
4. Women with Vulvodynia. -

Exclusion Criteria:

1. Women experiencing perimenopause or menopause.
2. Women with medical, or gynecological or hormonal abnormalities.
3. Women with mental disorders.
4. Women who use substances. -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Impact of Female Chronic Pelvic Pain Questionnaire (IF-CPPQ) | Up to 16 weeks
  Impact of Female Chronic Pelvic Pain Questionnaire (IF-CPPQ)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol